CLINICAL TRIAL: NCT03772509
Title: A Randomized Controlled Trial of Varying Introduction Mode to Improve Interactive Voice Response (IVR) Survey Performance in Bangladesh and Tanzania
Brief Title: Use of Introduction Mode to Improve Interactive Voice Response Surveys in Bangladesh and Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: The Bloomberg Family Foundation, Inc. (Other); Makerere University (Other); Institute of Epidemiology, Disease Control and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318-5
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2018-12

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; computer-assisted telephone interviews; introduction mode
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two introduction and consent modes: 1) computer-assisted telephone interviews, or 2) interactive voice response.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CATI (Experimental): Introduction and consent via computer assisted telephone interview
  Interventions: Other: CATI
- IVR (No Intervention): Introduction and consent via interactive voice response

INTERVENTIONS:
Other: CATI — The participants in this arm were read the introduction and asked for consent by a call center employee using computer-assisted telephone interviewing and then were sent a noncommunicable disease risk factor survey via interactive voice response. This mode was used to motivate participants to complete the survey.
  Arms: CATI

SUMMARY:
This study evaluates the effect of two different introduction modes on interactive voice response (IVR) survey cooperation, response, refusal, and contact rates, in Bangladesh and Tanzania.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling techniques, participants were randomized to one of two introduction modes, followed by a noncommunicable disease (NCD) risk factor survey. The two modes were computer assisted telephone interview (CATI), in which a call-center employee read the introduction to a participant and received oral consent from them, before sending them the NCD risk factor survey via IVR, or the entire survey, including the introduction and consent, being obtained via IVR. In IVR surveys, participants use their touch tone key pad to answer pre-recorded questions. (i.e. If you are male, press 1; If you are female, press 2). This study was conducted in both Bangladesh and Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Bangladesh, conversant in either English or Bangla language. In Uganda, conversant in either Luo, Luganda, Runyakitara, or English languages.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1511 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is complete interviews, P is partial interviews, and R is refusals and breakoffs.
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is refusals and breakoffs, I is complete interviews, P is partial interviews, and eU is the estimated eligible proportion of unknowns.
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, PhD, MBBS, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; George W. Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Institute of Epidemiology Disease Control and Research, Dhaka, Bangladesh
- Ifakara Health Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722